CLINICAL TRIAL: NCT02526888
Title: A Single-center, Open-label, Randomized, Two-way Crossover Study to Investigate the Effect of Multiple-dose Diltiazem on the Pharmacokinetics of a Single Dose of 25 mg ACT-541468 in Healthy Male Subjects
Brief Title: Pharmacokinetic Interaction Between Diltiazem and ACT-541468 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AC-078-103
Record Dates: First submitted 2015-08-14; First posted 2015-08-18 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Healthy Subjects
Keywords: pharmacokinetic; interaction
MeSH Terms: interventions — daridorexant; Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence AB (Experimental): During Period 1, subjects receive a single dose of ACT-541468 on Day 1. During Period 2, they receive Diltiazem from Day 1 to Day 7 and a single dose of ACT-541468 on Day 4
  Interventions: Drug: ACT-541468; Drug: Diltiazem
- Sequence BA (Experimental): During Period 1, subjects receive Diltiazem from Day 1 to Day 7 and a single dose of ACT-541468 on Day 4. During Period 2, they receive a single dose of ACT-541468 on Day 1
  Interventions: Drug: ACT-541468; Drug: Diltiazem

INTERVENTIONS:
Drug: ACT-541468 — Oral capsule (25 mg) as single dose
Drug: Diltiazem — Two oral capsules (2 x 120 mg) once daily from Day 1 to Day 7

SUMMARY:
The main objective of this study is to investigate whether repeated administration of a cardiac medication (diltiazem) can affect the pharmacokinetics (i.e., amount and time of presence in the blood) of ACT-541468

DETAILED DESCRIPTION:
Because ACT-541468 appears to be mainly metabolized by CYP3A4, it is deemed of interest to investigate the potential influence of diltiazem, a well-known CYP3A4 inhibitor on the pharmacokinetic profile of ACT-541468.

Safety of the concomitant administration of the two drugs will also be assessed

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Body mass index (BMI) between 18.0 and 28.0 kg/m2 (inclusive) at screening
* Healthy on the basis of physical examination,cardiovascular assessments and laboratory tests

Exclusion Criteria:

* Any contraindication to the study drugs
* History or presence of any disease or condition or treatment, which may put the subject at risk of participation in the study or may interfere with the absorption, distribution, metabolism or excretion of the study drugs
* History of narcolepsy or cataplexy or modified Swiss narcolepsy scale total score < 0
* Any circumstances or conditions, which, in the opinion of the investigator, may affect the subject's full participation in the study or compliance with the protocol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2015-11-01 (Actual); Study Completion 2015-11-01 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of ACT-541468 | From baseline to end of study (Day 8 after last study drug intake for sequence AB, Day 5 after last study drug intake for sequence BA)
  Cmax will be directly derived from the plasma concentration time curves of ACT-541468
Time to reach Cmax of ACT-541468 in plasma | From baseline to end of study (Day 8 after last study drug intake for sequence AB, Day 5 after last study drug intake for sequence BA
  tmax will be directly derived from the plasma concentration time curves of ACT-541468
Area under the plasma concentration-time curve (AUC) of ACT-541468 | From baseline to end of study (Day 8 after last study drug intake for sequence AB, Day 5 after last study drug intake for sequence BA)
  AUC will be calculated for the following time frame: from time zero to the last measured concentration above the limit of quantification and from time zero to infinitiy

OTHER OUTCOMES:
Incidence of safety events of interest | From baseline to end of study (Day 8 after last study drug intake for sequence AB, Day 5 after last study drug intake for sequence BA)
  Events of interest are any abnormalities in ECG, vital signs or laboratory test results
Incidence of adverse events | From baseline to end of study (Day 8 after last study drug intake for sequence AB, Day 5 after last study drug intake for sequence BA)
  Number of participants with any adverse events, including laboratory abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Laure Boof, PhD, Study Director — Actelion
Locations (1):
- CRS Clinical Research Services Kiel GmbH, Kiel, Germany